CLINICAL TRIAL: NCT05088317
Title: The Relationship of Exercise Capacity With Physical Activity Level, Sleep Apnea Risk and Quality of Life in Obese Adults
Brief Title: Relationship of Exercise Capacity With Physical Activity Level, Sleep Apnea Risk and Quality of Life in Obese Adults
Status: Completed | Type: Observational
Sponsor: Goksen Kuran Aslan (Other)
Responsible Party: Sponsor-Investigator, Goksen Kuran Aslan, Assoc. Prof. Goksen Kuran Aslan, Istanbul University
Organization: Istanbul University (Other)
Other Study IDs: 2021-31
Record Dates: First submitted 2021-09-24; First posted 2021-10-21 (Actual); Last update posted 2023-08-16 (Actual); Status verified 2023-08

CONDITIONS: Obesity
Keywords: obesity; exercise capacity; physical activity; sleep apnea; quality of life; anxiety; depression; hand grip strength
MeSH Terms: conditions — Obesity; Motor Activity; Sleep Apnea Syndromes; Anxiety Disorders; Depression

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Obese group: Volunteer female and male individuals aged 20-65 years, followed in an Internal Diseases unit of a state hospital in Turkey, diagnosed with obesity (BMI> 30 kg/m^2), who met the inclusion criteria of the study.
  Interventions: Diagnostic Test: Exercise capacity
- Healthy group: Healthy male and female individuals between the ages of 20-65 who were not diagnosed with obesity and volunteered to participate in the study.
  Interventions: Diagnostic Test: Exercise capacity

INTERVENTIONS:
Diagnostic Test: Exercise capacity — The incremental shuttle walking test at increasing speed (ISWT) is one of the field tests used to evaluate exercise capacity. It has been shown that ISWT is a valid and reliable assessment tool that can be used to evaluate exercise capacity in obese individuals. This test is an exercise test in which walking between two cones 10 m apart at increasing speed for 12 minutes is counted as one sit-up for each 10-meter walk between the two cones. It is continued until the patient is unable to continue the test due to shortness of breath, the heart rate reaches 85% of the maximum expected heart rate, or completes the 12-minute test. In this test, the primary measure is the distance walked, and the result is calculated based on the number of shuttles completed.

SUMMARY:
Volunteer female and male individuals aged 20-65 years, followed in the State Hospital Internal Diseases Unit, diagnosed with obesity (BMI> 30 kg/m^2), and meeting the inclusion criteria will be included in the study. The control group will consist of healthy male and female individuals between the ages of 20-65 who have not been diagnosed with obesity. The demographic and clinical characteristics of the participants who voluntarily accepted to participate in the study will be questioned with the "Evaluation Form" prepared by the researchers, and the body compositions of the participants will be evaluated. The "Charlson Comorbidity Index (CCI)" will be used to determine the existing chronic diseases of the participants and to evaluate participants' comorbidities. Next; the "Incremental Shuttle Walk Test (ISWT)" will be applied to determine exercise capacity. In addition, in order to determine the level of physical activity, a "pedometer" device will be given to the participants, participants will be asked to carry the device on them for 7 days, and at the end of the period, the pedometer data will be recorded. At the same time, participants will be required to fill in the "International Physical Activity Questionnaire-Short Form (IPAQ-SF)". Participants will be asked to fill in the "Stop-Bang Test" to assess the risk of sleep apnea, the "Obesity-Specific Quality of Life Scale (OSQOL)" to assess the health-related quality of life, and the "Hospital Anxiety and Depression Scale (HADS)" to determine the anxiety and depression level of the participants. Handgrip strength will be evaluated with a hydraulic hand dynamometer. Assessments take an average of 45 minutes is planned.

DETAILED DESCRIPTION:
Obesity is a serious public health problem whose prevalence is increasing day by day and is accepted as an epidemic by the World Health Organization. Obesity; increases the risk of developing cardiovascular and metabolic disorders such as atherosclerosis, type II diabetes and metabolic syndrome, but also leads to some types of cancer and many musculoskeletal disorders. In addition to all these negative diseases and syndromes, obese individuals often experience a significant deterioration in their physical functions. At the same time, the sedentary lifestyle, which is common in obese individuals, causes a decrease in exercise capacity, which negatively affects the ability to perform activities of daily living. Studies have shown that decreased exercise capacity is strongly correlated with the risk of all-cause mortality. In addition, patients with low exercise capacity have a higher risk of regaining the lost weight. Therefore, increasing exercise capacity is an important goal in obesity management as well as reducing body weight. Studies show that obese individuals are generally at risk for low physical activity levels, sleep apnea syndrome and low quality of life. On the other hand, there is not enough information about the relationship between exercise capacity, physical activity level, sleep apnea risk and quality of life in obese adults. Exercise capacity; investigation of its relationship with physical activity level, sleep apnea risk and quality of life will give an idea about the effect of exercise on these parameters if exercise capacity is increased with a comprehensive exercise program to be prepared for obese individuals. In conclusion, the aim of the study was to evaluate exercise capacity in obese adults and to investigate the relationship between exercise capacity, physical activity level, sleep apnea risk and quality of life.

ELIGIBILITY:
Inclusion criteria for obese participants:

* Between the ages of 20-65
* With BMI>30 kg/m^2

Inclusion criteria for healthy participants:

* Between the ages of 20-65
* With BMI<30 kg/m^2

Exclusion Criteria:

* Pregnancy
* Uncontrollable hypertension
* Uncontrolled diabetes requires the use of insulin
* Chronic lung diseases (COPD, etc.)
* Heart failure
* Cognitive and motor disorders
* Orthopedic and neurological dysfunctions that may interfere with evaluation

Ages: 20 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The obese population will consist of participants diagnosed with obesity (BMI> 30 kg/m^2), followed by the Tuzla State Hospital Internal Diseases unit in the Tuzla district of Istanbul. The healthy participant population will consist of healthy male and female individuals residing in Istanbul, between the ages of 20 and 65, who have not been diagnosed with obesity.
Sampling Method: Non-Probability Sample
Enrollment: 64 (Actual)
Dates: Start 2021-09-04 (Actual); Primary Completion 2022-09-04 (Actual); Study Completion 2022-12-04 (Actual)

PRIMARY OUTCOMES:
The Incremental Shuttle Walk Test | Baseline
  The incremental shuttle walking test at increasing speed is one of the field tests used to evaluate exercise capacity. This test is an exercise test in which walking between two cones 10 m apart at increasing speed for 12 minutes is counted as one sit-up for each 10-meter walk between the two cones. It is continued until the patient is unable to continue the test due to shortness of breath, the heart rate reaches 85% of the maximum expected heart rate, or completes the 12-minute test. In this test, the primary measure is the distance walked, and the result is calculated based on the number of shuttles completed.
Pedometer | The pedometer will be given to the participants on the day the participants are evaluated and it will be taken back after 7 days. At the end of 7 days, the total number of steps will be recorded.
  The pedometer is a cost-effective, easy-to-understand device that is usually worn on the waist with an apparatus, which allows to objectively evaluate the level of physical activity, measures the number of steps.
International Physical Activity Questionnaire-Short Form | Baseline
  It is a questionnaire used to record the duration of physical activity at different levels in the last week.
Stop-Bang Test | Baseline
  The Stop-Bang Test is one of the screening tests used to evaluate the risk of obstructive sleep apnea.
Obese-Specific Quality of Life Scale | Baseline
  Obese-Specific Quality of Life Scale: The scale consists of 17 items and is a six-point Likert type. The scale is reverse scored and the total score is 102. When the total score approaches zero, it indicates that the quality of life of the individuals decreases, and when it approaches 100, the quality of life increases.

SECONDARY OUTCOMES:
Hospital Anxiety and Depression Scale | Baseline
  7 items of the scale assess anxiety and 7 items assess depression. The answers, which are evaluated in a three-point Likert format, are scored between 0-3. When patients scored 0-10 for anxiety, patients were defined as no anxiety, 11 or more anxiety, and 0-7 points for depression as no depression, 8 or more depression.
Hydraulic Hand Dynamometer | Baseline
  Hydraulic Hand Dynamometer provides readings of grip strength.

CONTACTS AND LOCATIONS:
Locations (1):
- Istanbul University-Cerrahpasa, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No